CLINICAL TRIAL: NCT01793285
Title: Retrospective, Multicentric, National, Observational Study, to Follow-up the Patients Who Participated in the Loadet Study (RELOADET Study)
Brief Title: An Observational, Retrospective, Multicenter, National Study for the Monitoring of Subjects Who Participated in the LoadET Clinical Trial
Acronym: RELOADET
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801136; RELOADET
Record Dates: First submitted 2013-01-30; First posted 2013-02-15 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ETANERCEPT — During the LoadET study (0881A3-102090), subjects were treated with etanercept 100 mg versus 50 mg weekly. After completing this study, the subjects were allowed to continue the treatment with etanercept 50 mg weekly, etanercept 100 mg weekly, another drug, or abandoned medication at the discretion of their physician.
  This is a non-interventional study in which historic data will be collected retrospectively from the patient's clinical history. During the historical period covered in the Study, patients would have received the treatment and the medical care that their treating physicians considered appropriate under the conditions of standard clinical practice.

SUMMARY:
Previous studies suggest that an increase in doses of weekly etanercept from 50 mg to 100 mg improves the efficacy of the treatment in patients with cutaneous psoriasis, rheumatoid arthritis, and psoriatic arthritis. In this same line of study, during the 2007 2008 period, we conducted a multicenter, double-blind, 12-week Study (LoadET, 0881A3-102090) comparing the efficacy of etanercept at a standard dose (50 mg/week) versus a double dose (100 mg/week) in subjects with AS refractory to conventional therapy. The interim results of said study do not appear to support the value of doubling the dose of etanercept in the treatment of subjects with AS. Once this study was finalised, the subjects continued to be monitored by their regular physician, who decided on the dose and treatment to follow according to the conditions of standard clinical practice.

The objective of this observational study is to evaluate the course of the disease in the long-term (three years) under the conditions of standard clinical practice, in subjects who had participated in the LoadET study. Therefore, we would like to follow-up on those patients by reviewing their clinical histories for the three-year period between the finalisation of their participation in the LoadET Study (0881A3-102090) and now. This will allow us to assess the efficacy and survival of the drug, as well as the possible appearance of side effects in the three years following the finalisation of the study by comparing the results according to if the subjects had received 50 mg/week or 100 mg/week during the LoadET study (0881A3 102090).

DETAILED DESCRIPTION:
Given that this is a follow-up study of subjects who participated in the LoadET study (0881A3-102090), we have planned the inclusion of all subjects who completed said study, that is, 97 of the 108 subjects in the LoadET study.

ELIGIBILITY:
Inclusion Criteria:

* AS patients who had previously participated in the LoadET study (0881A3-102090).
* Subjects who completed the LoadET Study.
* Patients who grant their informed consent

Exclusion Criteria:

* Patients who participated in the LoadET study but who discontinued treatment and, therefore, did not complete the study.
* Patients without standard follow-up by the physician since the end of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ankylosing Spondylitis subjects who were treated with ETN when participating in the previous LoadET study (0881A3-102090)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Spain (13):
  - Pfizer Investigational Site, Madrid, Alcorcón
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Murcia, El Palmar
  - Pfizer Investigational Site, Barcelona, Hospitalet de Llobregat
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Madrid, Majadahonda
  - Pfizer Investigational Site, A Coruña
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Córdoba
  - Pfizer Investigational Site, Oviedo
  - Pfizer Investigational Site, Pamplona_Iruña_
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Valencia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801136&StudyName=An%20Observational%2C%20Retrospective%2C%20Multicenter%2C%20National%20Study%20for%20the%20Monitoring%20of%20Subjects%20Who%20Participated%20in%20the%20LoadET%20Clinical%20Tr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the LoadET study 0881A3-102090 (NCT00873730), were eligible for this study.
Groups:
- Etanercept: Participants who completed LoadET study 0881A3-102090 (NCT00873730) and received either etanercept 50 milligram (mg) weekly subcutaneously, etanercept 100 mg weekly subcutaneously, another drug, or abandoned medication as per standard clinical practice were observed retrospectively for 3 years.
Period: Overall Study
Arm/Group | Etanercept
Started | 85
Completed | 85
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Etanercept: Participants who completed LoadET study 0881A3-102090 (NCT00873730) and received either etanercept 50 mg weekly subcutaneously, etanercept 100 mg weekly subcutaneously, another drug, or abandoned medication as per standard clinical practice were observed retrospectively for 3 years.
Arm/Group | Etanercept
Number analyzed (Participants) | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 45.90 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Discontinued Treatment With Etanercept
Description: Participants who discontinued etanercept following 3 years after finalization of LoadET study 0881A3-102090 (NCT00873730) due to any of these reason were reported: adverse events, failure in therapeutic response, disease remission and discontinued for other causes.
Time Frame: Baseline up to Year 3
Population: Analysis population included all participants who had previously participated in the LoadET study (NCT00873730) and fulfilled all the eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 85
percentage of participants | 41.2

2. Secondary Outcome: Time Between the Onset of Ankylosing Spondylitis Symptoms and First Visit to the Rheumatologist
Description: Time passed since the ankylosing spondylitis symptoms started until the participant arrived for the first time to visit the rheumatologist was reported. Ankylosing spondylitis symptoms may include pain, stiffness, axial manifestations, and enthesitis etc.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Etanercept
Number analyzed (Participants) | 85
years | 6.35 (7.27)

3. Secondary Outcome: Time to Diagnosis of Ankylosing Spondylitis
Description: Time to first diagnosis of alkylosing spondylitis was reported.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Etanercept
Number analyzed (Participants) | 85
years | 7.53 (8.01)

4. Secondary Outcome: Number of Participants Who Received Non-pharmacological Treatment
Description: Participants who received any non-pharmacological treatment (participant education, regular exercises and physical therapy) in the 3 years since the last LoadET study 0881A3-102090 (NCT00873730) visit were reported.
Time Frame: Baseline up to Year 3
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 85
participants | 3

5. Secondary Outcome: Number of Participants Who Received Pharmacological Treatment
Description: Participants who received any pharmacological treatment (non-steroidal anti-inflammatory drugs [NSAIDs], disease-modifying antirheumatic drugs [DMARDs], corticosteroids and other treatments including anti-tumor necrosis factor-alpha [TNFalpha] or other biological agents etc.) in the 3 years since the last LoadET study 0881A3-102090 (NCT00873730) visit were reported.
Time Frame: Baseline up to Year 3
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 85
participants
  NSAIDs | 55
  DMARDs | 15
  Corticosteroids | 7
  Other | 26

6. Secondary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score
Description: Participants disease activity assessed using a 100 millimeter (mm) Visual Analog Scale (VAS), ranging from 0 = very good to 100 = very bad.
Time Frame: Baseline, Year 1, 2, 3
Population: Analysis population included all evaluable participants who continued the treatment at 3 years after the finalizing of the LoadET study (0881A3-102090). Here, N (number of participants analyzed) signifies those participants who were evaluable for this measure. n=number of participants evaluable for this measure at specified time point.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 49
mm
  Baseline (n=43) | 1.70 [0.80 to 3.70]
  Year 1 (n=33) | 2.00 [0.20 to 4.00]
  Year 2 (n=32) | 2.00 [1.00 to 3.00]
  Year 3 (n=49) | 1.40 [0.90 to 3.00]

7. Secondary Outcome: Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: BASFI is a validated self-assessment tool that determines the degree of functional limitation in ankylosing spondylitis. Utilizing a VAS of 0-10, 0 = easy, 10 = impossible, participants answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a sum of the scores of the 10 questions, final score ranged from 0-100, where higher score referred to higher impairment in the functional ability.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 48
units on a scale
  Baseline (n=45) | 26.00 [8.90 to 47.00]
  Year 1 (n=30) | 23.10 [8.00 to 43.50]
  Year 2 (n=25) | 23.00 [10.00 to 42.50]
  Year 3 (n=48) | 24.05 [13.05 to 35.80]

8. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participant with ankylosing spondylitis. Utilizing a VAS of 0-10, 0=none and 10=very severe participant's answered 6 questions measuring discomfort, pain and fatigue. The final BASDAI score is a sum of the individual assessments. Final score ranged from 0-60, higher score indicates higher disease activity.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 48
units on a scale
  Baseline (n=45) | 9.90 [5.30 to 21.00]
  Year 1 (n=34) | 10.60 [4.00 to 16.70]
  Year 2 (n=28) | 10.50 [5.05 to 17.10]
  Year 3 (n=48) | 9.30 [4.09 to 17.25]

9. Secondary Outcome: Spinal Pain as Assessed Using Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: Participant's spinal pain - was assessed by answering question 2 of BASDAI on a 0 to10 VAS; participants were asked: "How would you describe the overall level of ankylosing spondylitis neck, back or hip pain you have had?" 0 =none and 10 =very severe.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 48
units on a scale
  Baseline (n=45) | 2.20 [0.80 to 5.20]
  Year 1 (n=33) | 2.90 [1.00 to 4.40]
  Year 2 (n=27) | 3.00 [1.00 to 4.30]
  Year 3 (n=48) | 2.00 [0.75 to 4.00]

10. Secondary Outcome: Fatigue as Assessed Using Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: Participant's fatigue was assessed by answering question 1 of BASDAI on a 0 to 10 VAS; participants were asked: "How would you describe the overall level of fatigue/tiredness you have experienced?" 0=none and 10=very severe.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 48
units on a scale
  Baseline (n=45) | 1.70 [0.80 to 5.00]
  Year 1 (n=33) | 2.00 [0.60 to 4.10]
  Year 2 (n=27) | 1.50 [1.00 to 3.00]
  Year 3 (n=48) | 2.00 [0.90 to 4.00]

11. Secondary Outcome: Modified Schober's Test
Description: Measurement in centimeters (cm) of the distance between marks originally placed while the participant was standing erect 10 cm above and 5 cm below the midpoint of a line that joints the posterior superior iliac spines. Distance between marks was re-measured (in cm rounded to the nearest 0.1 cm) with participant maximally bend forward, knees fully extended, with spine in full flexion. The measurement of two attempts was made.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 44
cm
  Baseline (n=43) | 17.75 [4.65 to 20.00]
  Year 1 (n=25) | 13.00 [5.50 to 18.80]
  Year 2 (n=25) | 11.00 [5.00 to 18.00]
  Year 3 (n=44) | 15.45 [4.75 to 19.13]

12. Secondary Outcome: Occiput-to-wall Distance
Description: Occiput-to-wall distance: distance between the occiput (posterior or back portion of the head) and the wall when the participant stood with heels and shoulder against the wall and the back straight. The distance between the occiput and the wall was measured in cm (rounded to the nearest 0.1 cm), in two attempts.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 45
cm
  Baseline (n=43) | 0.00 [0.00 to 8.50]
  Year 1 (n=25) | 0.00 [0.00 to 8.00]
  Year 2 (n=22) | 2.00 [0.00 to 9.00]
  Year 3 (n=45) | 0.00 [0.00 to 3.50]

13. Secondary Outcome: Chest Expansion Measurement
Description: Chest expansion, measured in cm (rounded to the nearest 0.1 cm), is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line). Chest expansion was measured for both maximum and minimum inhalation. The measurement of two attempts was made.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 39
cm
  Baseline: Maximum Inspiration (n=39) | 98.00 [86.25 to 106.00]
  Baseline: Minimum Inspiration (n=32) | 98.13 [88.25 to 105.50]
  Year 1: Maximum Inspiration (n=5) | 96.25 [86.75 to 108.00]
  Year 1: Minimum Inspiration (n=5) | 101.00 [80.75 to 104.50]
  Year 2: Maximum Inspiration (n=6) | 100.50 [82.00 to 113.00]
  Year 2: Minimum Inspiration (n=7) | 86.00 [8.00 to 109.00]
  Year 3: Maximum Inspiration (n=36) | 96.75 [85.75 to 106.50]
  Year 3: Minimum Inspiration (n=32) | 94.38 [86.63 to 104.00]

14. Secondary Outcome: C-reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: milligram per milliliter (mg/mL)
Arm/Group | Etanercept
Number analyzed (Participants) | 49
milligram per milliliter (mg/mL)
  Baseline (n=45) | 0.27 [0.10 to 0.84]
  Year 1 (n=46) | 0.25 [0.10 to 0.82]
  Year 2 (n=47) | 0.47 [0.16 to 0.95]
  Year 3 (n=49) | 0.40 [0.18 to 1.19]

15. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter/hour (mm/hr). A higher rate is consistent with inflammation.
Time Frame: Baseline, Year 1, 2, 3
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: mm/hr
Arm/Group | Etanercept
Number analyzed (Participants) | 50
mm/hr
  Baseline (n=50) | 2.00 [2.00 to 7.00]
  Year 1 (n=44) | 4.00 [2.00 to 7.50]
  Year 2 (n=49) | 4.00 [2.00 to 8.00]
  Year 3 (n=46) | 6.00 [3.00 to 11.00]

16. Secondary Outcome: Lipid Profile: Total Cholesterol (TC), High Density Lipoprotein (HDL) and Triglycerides Levels
Description: Lipid profile included following parameters: Total Cholesterol (TC), high-density lipoprotein (HDL) and triglycerides (TGs).
Time Frame: Baseline, Year 1, 2, 3
Population: Analysis population included all evaluable participants who continued the treatment at 3 years after the finalizing of the LoadET study (0881A3-102090). Here, N (number of participants analyzed) signifies those participants who were evaluable for this measure. n=number of participants evaluable for each parameter at specified time point.
Measure: Median (Inter-Quartile Range); unit: milligram per deciliter (mg/dL)
Arm/Group | Etanercept
Number analyzed (Participants) | 42
milligram per deciliter (mg/dL)
  Baseline: Total Cholesterol (n=42) | 189.50 [167.00 to 210.00]
  Baseline: High Density Lipoprotein (n=18) | 53.00 [45.00 to 59.00]
  Baseline: Triglycerides (n=34) | 77.00 [61.00 to 113.00]
  Year 1: Total Cholesterol (n=35) | 191.00 [170.00 to 210.00]
  Year 1: High Density Lipoprotein (n=24) | 58.00 [47.50 to 66.00]
  Year 1: Triglycerides (n=32) | 89.50 [73.00 to 147.00]
  Year 2: Total Cholesterol (n=39) | 191.00 [166.00 to 209.00]
  Year 2: High Density Lipoprotein (n=28) | 57.00 [45.00 to 64.50]
  Year 2: Triglycerides (n=34) | 103.50 [72.00 to 134.00]
  Year 3: Total Cholesterol (n=40) | 184.00 [172.00 to 205.50]
  Year 3: High Density Lipoprotein (n=23) | 51.00 [43.00 to 59.00]
  Year 3: Triglycerides (n=32) | 102.50 [79.00 to 124.00]

17. Secondary Outcome: Time to Treatment Discontinuation With Etanercept
Description: Time to treatment discontinuation with etanercept was assessed retrospectively at Year 3 for participants who did not discontinue treatment at the end of previous LoadET study 0881A3-102090 (NCT00873730). It was defined as time from first dose of etanercept received in the previous LoadET study 0881A3-102090 (NCT00873730) to last dose of etanercept.
Time Frame: Year 3
Population: Analysis population included all evaluable participants who continued the treatment at 3 years after the finalizing of the LoadET study (0881A3-102090). Here, N (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (95% Confidence Interval); unit: years
Arm/Group | Etanercept
Number analyzed (Participants) | 78
years | 3.56 [3.20 to 3.91]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 2/85
Other Adverse Events (participants affected / at risk) | 31/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=85)
Cronhn's disease (Gastrointestinal disorders) | 1
Cholesystectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=85)
Treatment failure (General disorders) | 10
Dizziness (Nervous system disorders) | 6
Uveitis (Eye disorders) | 5
Respiratory tract infection (Infections and infestations) | 3
Iridocyclitis (Eye disorders) | 3
Chickenpox (Infections and infestations) | 2
Renal colic (Renal and urinary disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Headache (Nervous system disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 2
Epicondylitis (Injury, poisoning and procedural complications) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Surgery (Surgical and medical procedures) | 1
Sinus tachycardia (Cardiac disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
Pharyngitis (Infections and infestations) | 1
Pain (General disorders) | 1
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1
Oesophageal spasm (Gastrointestinal disorders) | 1
Muscle tension (Musculoskeletal and connective tissue disorders) | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Gingival abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Episcleritis (Eye disorders) | 1
Epididymitis (Reproductive system and breast disorders) | 1
Oedema administration (General disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Bronchitis (Infections and infestations) | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1
Balanitis (Reproductive system and breast disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Acute sinusitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.